CLINICAL TRIAL: NCT01701674
Title: Co-stimulation With Ipilimumab to Enhance Lymphodepletion Plus Adoptive Cell Transfer and High Dose IL-2 in Patients With Metastatic Melanoma
Brief Title: Ipilimumab With Lymphodepletion Plus Adoptive Cell Transfer and High Dose IL-2 in Melanoma Mets Pts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry); Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17057; CA184-213 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Melanoma
Keywords: skin cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Ipilimumab; Cyclophosphamide; fludarabine; fludarabine phosphate; Interleukin-2; aldesleukin; Toll-Like Receptor 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combination Therapy (Experimental): The combination of ipilimumab followed by lymphodepletion with chemotherapy, TIL infusion, and high dose IL-2.
  Interventions: Drug: Ipilimumab; Procedure: Tumor Infiltrating Lymphocytes (TIL); Drug: Administration of Lymphodepletion; Drug: Cyclophosphamide as Part of Lymphodepletion; Drug: Fludarabine as Part of Lymphodepletion; Drug: High Dose IL-2; Biological: Adoptive Cell Therapy with TIL

INTERVENTIONS:
Drug: Ipilimumab — Pre-treatment with ipilimumab (cycle 1): Before the participant's tumor sample is taken to send to the lab for growing the TILs, they will start their first cycle of ipilimumab. This drug is given as an intravenous infusion (through a vein) over a period of about 90 minutes (an hour and a half). Cycle 2 of ipilimumab: About a week after the sample of the participant's tumor was collected for TIL growth (and 3 weeks after their first cycle of ipilimumab), participants will have their second cycle of ipilimumab. This will be another IV infusion, lasting about 90 minutes.
  Other Names: Yervoy
Procedure: Tumor Infiltrating Lymphocytes (TIL) — Tumor sample for TIL growth in the lab: About 2 weeks after the participant's first cycle of ipilimumab, a sample of their tumor will be collected and sent to the lab for TIL growth. Growing the TILs takes about 6 weeks. If their sample has grown enough TIL cells, participants will continue with the next part of the study. Depending on how long the TILs take to grow in the lab, they may need to repeat some of their laboratory and imaging tests (blood draws, X-rays, and CT or magnetic resonance imaging [MRI] scans). TIL Infusion (inpatient): After completing lymphodepletion, participants will be admitted back into the hospital for IV infusion of the TIL cells.
Drug: Administration of Lymphodepletion — Lymphodepletion (inpatient hospital stay for about 2 days plus outpatient drug dosing for 5 days): About 4 weeks after their second cycle of ipilimumab, participants will be admitted to the hospital for their first two days of receiving the chemotherapy drug, cyclophosphamide. This drug will be given as an intravenous (IV, meaning through the vein) infusion. After 2 days of receiving cyclophosphamide, if their study doctor thinks that they are well enough, you will be discharged from the hospital and will return for the next 5 days in a row for outpatient IV infusions of the second lymphodepletion chemotherapy, fludarabine.
Drug: Cyclophosphamide as Part of Lymphodepletion
  Other Names: Cytoxan
Drug: Fludarabine as Part of Lymphodepletion
  Other Names: Fludara
Drug: High Dose IL-2 — High dose IL-2 (continued inpatient): Participants will remain in the hospital following TIL infusion for receiving high dose IL-2 and recovery. The IL-2 will be given three times per day for about 3-5 days as an IV bolus (meaning through the vein, more quickly than other infusions - in about 15 minutes each dose). Participants will remain in the hospital for approximately 7-14 days until they have recovered from the IL-2 treatments.
  Other Names: Interleukin-2; Aldesleukin; Proleukin
Biological: Adoptive Cell Therapy with TIL
  Other Names: ACT

SUMMARY:
Purpose of this Pilot Study: The investigators want to study the safety, side effects, and benefits of tumor infiltrating lymphocytes (TILs), when they are given with the drug ipilimumab. Ipilimumab is a type of immunotherapy - a drug that is used to boost the ability of the immune system to fight cancer, infection, and other diseases.

DETAILED DESCRIPTION:
The primary endpoints of this pilot trial will be the safety and feasibility of administering ipilimumab with Adoptive Cell Therapy (ACT) using TIL. The data analysis will mainly be descriptive. All study results will be preliminary and of exploratory in nature due to the pilot status and small sample size of the trial. Feasibility is defined as the ability to deliver at least 50% (i.e., two out of four) of the planned doses of ipilimumab and successfully treat at least 60% (i.e., ≥ 6/10) of the patients with TIL. All participants will be evaluable for toxicity from the time of their first protocol treatment. Toxicity will be reported by type and severity according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) version 4.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have unresectable metastatic stage IV melanoma or stage III intransit or regional nodal disease, and in the opinion of the institutional PI is an acceptable candidate for ACT with high dose IL-2
* Residual measurable disease after resection of target lesion(s) for TIL growth
* Tumor may have a B-RAF V600 mutation or be BRAF wild type, and patients must not have been previously treated with ipilimumab
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 - 1. ECOG performance status of 0-1 will be inferred if the patient's level of energy is ≥ 50% of baseline.
* May have been previously treated for metastatic disease, or may have not had prior systemic treatment. Patients with a V600 BRAF mutated tumor may have previously received a prior BRAF inhibitor.
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of screening.
* Adequate renal, hepatic and hematologic function, including creatinine of less than or equal to 1.7 gm/dL, total bilirubin less than or equal to 2.0 mg/dL, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dL, aspartate aminotransferase (AST) and alanine transaminase (ALT) of less than 3 X institutional upper limit of normal, hemoglobin of 8 gm/dL or more, white blood count (WBC) of 3000 per mcL and total granulocytes of 1000 per mcL or more, and platelets of 100,000 per mcL or more.
* Must have a positive screening Epstein-Barr virus (EBV) antibody titre on screening test
* Potential participants with antibiotic allergies per se are not excluded; although the production of TIL for adoptive transfer includes antibiotics, extensive washing after harvest will minimize systemic exposure to antibiotics.
* At screening, patients with ≤ 3 untreated CNS metastases may be included provided none of the untreated lesions are > 1 cm in greatest dimension, and there is no peri-tumoral edema present on brain imaging (MRI or CT if MRI is contraindicated).
* At screening, patients with central nervous system (CNS) metastases treated with either surgical resection and/or radiation therapy may be included. Patients may be included if the largest lesion is ≤ 1 cm, and there is no evidence of progressive CNS disease on brain imaging at least 28 days after treatment.
* At screening, patients may be included if the largest lesion is > 1 cm or > 3 in number, and there is no evidence of progressive CNS disease on brain imaging at least 90 days after treatment with surgery and/or radiation therapy.
* No evidence of ongoing cardiac dysrhythmia ≥ grade 2 (NCI Common Terminology Criteria for Adverse Events [CTCAE], v4.0)
* All laboratory and imaging studies must be completed and satisfactory within 30 days of signing the consent document, with the exceptions of: negative serum pregnancy test for women of child-bearing potential which must be negative within 7 days of screening, human leukocyte antigen (HLA) typing which will not be repeated if performed previously, and pulmonary function tests (PFTs)/cardiac stress tests whose results are valid for 6 months if performed previously.

Exclusion Criteria:

* Active systemic infections requiring intravenous antibiotics, coagulation disorders or other major medical illness of the cardiovascular, respiratory or immune system, which in the opinion of the principal investigator (PI) or treating coinvestigator is not acceptable risk for ACT, are excluded.
* Testing positive for HIV titre, Hepatitis B surface antigen, Hepatitis B core antibody, Hepatitis C antibody, Human T-Lymphotropic Virus (HTLV) I or II antibody, or both Rapid. Plasma Reagin (RPR) and fluorescent treponemal antibodies (FTA) positive are excluded.
* Pregnant or nursing
* Patients needing chronic, immunosuppressive systemic steroids are excluded
* History of autoimmune disease that require immunosuppressive medications at the time of screening
* Presence of a significant psychiatric disease, which in the opinion of the principal investigator or his designee, would prevent adequate informed consent or render immunotherapy unsafe or contraindicated
* Patients with > 3 untreated CNS metastases or evidence of peri-tumoral edema
* Patients with ≤ 3 untreated CNS metastases but with at least one lesion >1 cm or peri-tumoral edema
* Patients with invasive malignancy other than melanoma at the time of enrollment and within 2 years prior to the first TIL administration are excluded, except for adequately treated (with curative intent) basal or squamous cell carcinoma, in situ carcinoma of the cervix, in situ ductal adenocarcinoma of the breast, in situ prostate cancer, or limited stage bladder cancer or other cancers from which the patient has been disease-free for at least 2 years.
* Patients with treated CNS metastases > 1 cm or > 3 in number will be excluded if there is evidence of progressive CNS disease on brain imaging at least 90 days after treatment with surgery and/or radiation therapy.
* Unable to comprehend and give informed consent
* Male patients with WOCBP partners who do not agree to use two FDA-accepted forms of contraception during sexual intercourse with women of child-bearing potential from the start of ipilimumab and up to at least 6 months after ACT
* WOCBP who do not agree to use 2 FDA forms of contraception during sexual intercourse from the start of ipilimumab and up to at least 6 months after ACT
* Patients who have received ipilimumab in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-10-09 (Actual); Primary Completion 2016-04-21 (Actual); Study Completion 2025-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amod Sarnaik, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center, April 2013 through July 2014.
Groups:
- Experimental: Combination Therapy: The combination of ipilimumab followed by lymphodepletion with chemotherapy, TIL infusion, and high dose IL-2.
Period: Overall Study
Arm/Group | Experimental: Combination Therapy
Started | 13
Completed | 12
Not Completed | 1
Not completed — Unable to safely complete treatment | 1

BASELINE CHARACTERISTICS:
Population: All participants (13). All evaluable participants (12) may be referenced for some outcome measures.
Arm/Group | Experimental: Combination Therapy
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 49 [22 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Dose Limiting Toxicity (DLT) Events
Description: Occurrence of adverse events with dose limiting toxicity, per adverse event category.
Time Frame: 3 months
Population: All participants
Measure: Number; unit: DLT events
Arm/Group | Experimental: Combination Therapy
Number analyzed (Participants) | 13
DLT events
  Eye-related: Uveitis | 1
  Gastrointestinal: Colitis | 1

2. Primary Outcome: Rate of Meeting Feasibility Requirements
Description: Number of participants who were successfully treated with at least 2 doses of ipilimumab and received TIL. Feasibility is defined as the ability to deliver at least 50% (i.e., two out of four) of the planned doses of ipilimumab and successfully treat at least 60% (i.e., ≥ 6/10) of the patients with TIL.
Time Frame: 3 months
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Combination Therapy
Number analyzed (Participants) | 13
Participants | 12

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response: Complete Response (CR) + Partial Response (PR), per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1 for target lesions and assessed by computed tomography (CT) scan. CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of the longest diameter (LD) of target lesions..
Time Frame: 12 weeks
Population: All participants.
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Combination Therapy
Number analyzed (Participants) | 13
percentage of participants | 38.5

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) per RECIST V1.1, defined as the time from study entry to disease progression, relapse or death due to any cause, whichever is earlier, will be summarized with the Kaplan-Meier curve. Progressive Disease (PD): At least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 42 months
Population: All participants.
Measure: Median (Full Range); unit: months
Arm/Group | Experimental: Combination Therapy
Number analyzed (Participants) | 13
months | 7.4 [1.5 to 42]

ADVERSE EVENTS:
Time Frame: 3 years, 6 months
Arm/Group | Experimental: Combination Therapy
Serious Adverse Events (participants affected / at risk) | 9/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Combination Therapy (N=13)
Hypothyroidism (Endocrine disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Autoimmune disorder (Immune system disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Investigations - Other, SIADH (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Cystitis non-infective (Renal and urinary disorders) | 2 (2)
Renal and urinary disorders - Other, Cistitis infective (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Combination Therapy (N=13)
Anemia (Blood and lymphatic system disorders) | 12 (82)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 (10)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 3 (4)
Palpitations (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 9 (12)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Endocrine disorders - Other (Endocrine disorders) | 3 (4)
Hypothyroidism (Endocrine disorders) | 1 (2)
Blurred vision (Eye disorders) | 3 (3)
Cataract (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 2 (2)
Eye disorders - Other (Eye disorders) | 3 (4)
Eye pain (Eye disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (8)
Bloating (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 7 (10)
Diarrhea (Gastrointestinal disorders) | 11 (30)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 5 (6)
Mucositis oral (Gastrointestinal disorders) | 4 (6)
Nausea (Gastrointestinal disorders) | 13 (31)
Vomiting (Gastrointestinal disorders) | 9 (11)
Chills (General disorders) | 10 (16)
Edema limbs (General disorders) | 5 (8)
Fatigue (General disorders) | 11 (33)
Fever (General disorders) | 7 (12)
Flu like symptoms (General disorders) | 3 (4)
General disorders and administration site conditions - Other (General disorders) | 7 (15)
Localized edema (General disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 7 (13)
Allergic reaction (Immune system disorders) | 1 (1)
Immune system disorders - Other (Immune system disorders) | 2 (2)
Bronchial infection (Infections and infestations) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 5 (5)
Mucosal infection (Infections and infestations) | 1 (1)
Penile infection (Infections and infestations) | 1 (2)
Upper respiratory infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Wound infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 3 (4)
Alanine aminotransferase increased (Investigations) | 11 (24)
Alkaline phosphatase increased (Investigations) | 9 (18)
Aspartate aminotransferase increased (Investigations) | 12 (26)
Blood bilirubin increased (Investigations) | 5 (11)
Cardiac troponin T increased (Investigations) | 1 (1)
CPK increased (Investigations) | 6 (9)
Creatinine increased (Investigations) | 3 (5)
INR increased (Investigations) | 1 (1)
Investigations - Other (Investigations) | 2 (7)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 12 (45)
Lymphocyte count increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 12 (32)
Platelet count decreased (Investigations) | 12 (61)
Serum amylase increased (Investigations) | 1 (1)
Weight gain (Investigations) | 1 (4)
White blood cell decreased (Investigations) | 12 (49)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 8 (10)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (7)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 12 (37)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (8)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (7)
Hyponatremia (Metabolism and nutrition disorders) | 10 (32)
Hypophosphatemia (Metabolism and nutrition disorders) | 12 (21)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Dizziness (Nervous system disorders) | 7 (10)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 10 (12)
Nervous system disorders - Other (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (4)
Acute kidney injury (Renal and urinary disorders) | 1 (2)
Bladder spasm (Renal and urinary disorders) | 1 (2)
Cystitis non-infective (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (4)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 1 (3)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (18)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (18)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (22)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 7 (9)
Surgical and medical procedures - Other (Surgical and medical procedures) | 2 (2)
Capillary leak syndrome (Vascular disorders) | 4 (4)
Flushing (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)
Hypotension (Vascular disorders) | 9 (14)
Lymphedema (Vascular disorders) | 3 (3)
Vascular disorders - Other (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes